CLINICAL TRIAL: NCT00001885
Title: Pulmonary Fibrosis Associated With Rheumatoid Arthritis: Identification of Genetic Polymorphisms
Brief Title: Identification of Genes Associated With Lung Disease in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990069; 99-H-0069
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: Healthy; Pulmonary Fibrosis; Rheumatoid Arthritis
Keywords: Interstitial Lung Disease; Inherited Disease; Genetic Markers; Alpha 1 Protease Inhibitor; DNA Mutations; Rheumatoid Arthritis; Pulmonary Fibrosis; Normal Volunteer
MeSH Terms: conditions — Pulmonary Fibrosis; Arthritis, Rheumatoid; Lung Diseases, Interstitial; Genetic Diseases, Inborn; alpha 1-Antitrypsin Deficiency

SUMMARY:
Pulmonary fibrosis (PF) is a condition in which the lungs of a patient become scarred and fibrous. It has been known to occur in as many as 40% of patients diagnosed with rheumatoid arthritis (RA). The cause of the pulmonary fibrosis in patients with RA is unknown.

Data gathered from previous research studies suggest that genetics may play a role in the development of PF in patients with rheumatoid arthritis. However, the actual genetic factors involved in the disease process have not been identified.

The goal of this study is to identify the genetic markers in patients with pulmonary fibrosis and rheumatoid arthritis.

DETAILED DESCRIPTION:
Pulmonary fibrosis that develops within a subpopulation of patients with rheumatoid arthritis is a disorder of unknown etiology. Although previous reports suggest that some individuals with rheumatoid arthritis have a genetic predisposition to the development of fibrotic lung disease, genetic factors have not been clearly identified. It is the intent of this clinical protocol to identify genetic polymorphisms in individuals with pulmonary fibrosis and rheumatoid arthritis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals 21 years of age or older with any of the following:

RA (based on 1987 American College of Rheumatology Revised Criteria for the Classification of RA) with PF (biopsy-proven), or

RA-only, or

Biopsy-proven idiopathic PF-only, or

Healthy research volunteers.

EXCLUSION CRITERIA:

Individuals with any of the following:

Inhalational exposure to fibrogenic fibers or dusts (e.g., asbestos, silica, coal, beryllium).

Chronic pulmonary disorders other than pulmonary fibrosis.

Other collagen vascular disorders (e.g., systemic lupus erythematosus, scleroderma, polymyositis, mixed connective tissue disease).

Non-rheumatoid arthritis.

Viral infections associated with PF (e.g., hepatitis B, hepatitis C, human immunodeficiency virus).

Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1999-03-21; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hakala M. Poor prognosis in patients with rheumatoid arthritis hospitalized for interstitial lung fibrosis. Chest. 1988 Jan;93(1):114-8. doi: 10.1378/chest.93.1.114. PMID 3335140